CLINICAL TRIAL: NCT01238341
Title: Prospective Evaluation of Clinical Utility of Endoscopic Retrograde Cholangiopancreatography (ERCP) With Overtube in Patients With Altered Gastric Anatomy
Brief Title: Evaluation of Pancreatobiliary Disorders in Patients With Altered Gastric Anatomy
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Pancreatobiliary disorders
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Pancreatobiliary Disease; Altered Gastric Anatomy
Keywords: Pancreatobiliary disease in patients with altered gastric anatomy.
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatobiliary disease: Patients who have altered gastric anatomy who need an ERCP with an overtube for evaluation of pancreatobiliary disease.
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangiopancreatography (ERCP) — An Endoscopic Retrograde Cholangiopancreatography (ERCP) performed with an overtube in the evaluation of pancreatobiliary disease in patients with altered gastric anatomy

SUMMARY:
In patients, who have altered gastric anatomy and pancreatobiliary disease, the use of an endoscopic overtube to facilitate an Endoscopic Retrograde Cholangiopancreatography (ERCP).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject has medical indication for Endoscopic Retrograde Cholangiopancreatography (ERCP)
3. Subject has altered gastric anatomy
4. Subject must be able to give informed consent.

Exclusion Criteria:

1. Any contraindication for Endoscopic Retrograde Cholangiopancreatography (ERCP) with overtube
2. The subject is unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a medical indication for ERCP and have altered gastric anatomy and are referred for the procedure as part of their standard medical care will be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2007-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Florida
Locations (1):
- Shands at UF Endoscoppy Center, Gainesville, Florida, United States

REFERENCES:
- [Derived] Wagh MS, Draganov PV. Prospective evaluation of spiral overtube-assisted ERCP in patients with surgically altered anatomy. Gastrointest Endosc. 2012 Aug;76(2):439-43. doi: 10.1016/j.gie.2012.04.444. No abstract available. PMID 22817798

RESULTS

PARTICIPANT FLOW:
Groups:
- Altered Gastric Anatomy: Patients with altered gastric anatomy that needed an Endoscopic Retrograde Cholangiopancreatography (ERCP) for endoscopic therapy of pancreatobiliary disease underwent ERCP with spiral overtube assisted enteroscopy.
Period: Overall Study
Arm/Group | Altered Gastric Anatomy
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Altered Gastric Anatomy
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 59.3 [39 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 7
Postsurgical anatomy [Number; unit: participants]
  Roux-en-Y hepaticojejunostomy | 2
  Roux-en-Y gastric bypass | 3
  Roux-en-Y gastric bypass with hepaticojejunostomy | 1
  Billroth II gastrectomy w/ Braun enteroenterostomy | 1
Indications for Endoscopic Retrograde Cholangiopancreatography (ERCP) [Number; unit: participants]
  Biliary obstruction | 5
  Bile duct stones | 1
  Pancreatic leak | 1

OUTCOME MEASURES:

1. Primary Outcome: Papilla or Duct-enterostomy Was Reached
Time Frame: During procedure, up to 3 hours
Measure: Number; unit: ERCPs
Units Other Than Participants: ERCP attempts
Arm/Group | Altered Gastric Anatomy
Number analyzed (Participants) | 7
Number analyzed (ERCP attempts) | 13
ERCPs | 10

2. Secondary Outcome: Successful Cannulation of the Duct of Intent
Description: Deep cannulation of the bile/pancreatic duct was indicated in 12 of 13 ERCPs, one procedure was performed for stent removal only. This outcome was only relevant when deep cannulation was clinically indicated, therefore this outcome was determined out of 12 ERCPs.
Time Frame: During procedure, up to 3 hours
Measure: Number; unit: ERCPs
Units Other Than Participants: ERCPs
Arm/Group | Altered Gastric Anatomy
Number analyzed (Participants) | 7
Number analyzed (ERCPs) | 12
ERCPs | 8

3. Secondary Outcome: Successful Endoscopic Therapy
Time Frame: During procedure, up to 3 hours
Measure: Number; unit: ERCPs
Units Other Than Participants: ERCPs
Arm/Group | Altered Gastric Anatomy
Number analyzed (Participants) | 7
Number analyzed (ERCPs) | 13
ERCPs | 9

4. Secondary Outcome: Total Procedure Time
Time Frame: During procedure, up to 3 hours
Measure: Mean (Full Range); unit: minutes
Units Other Than Participants: ERCPs
Arm/Group | Altered Gastric Anatomy
Number analyzed (Participants) | 7
Number analyzed (ERCPs) | 13
minutes | 95.6 [24 to 149]

ADVERSE EVENTS:
Arm/Group | Altered Gastric Anatomy
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes